CLINICAL TRIAL: NCT00798200
Title: CanWell: YMCA Based Exercise Program for Well Cancer Survivors
Brief Title: Community Based Exercise Program for Well Cancer Survivors
Acronym: CanWell
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Oren Cheifetz, Clinical Specialist - Physiotherapy, Hamilton Health Sciences Corporation
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: WorkForceOntario 001
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
Keywords: Cancer; Oncology; Rehabilitation; Endurance; Strength
MeSH Terms: conditions — Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Other): All participants will take part in a supervised, structured, exercise program
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — All exercise programs will include endurance and strength exercises.

SUMMARY:
This project will create a community based exercise program for well cancer survivors. The goal is that the YMCA will gain the competence to work with this unique population in a safe and productive manner.

DETAILED DESCRIPTION:
All well, adult, cancer survivors are eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* All well cancer survivors who are medically stable.

Exclusion Criteria:

* Children are not eligible for this project.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Endurance measure (STEEP treadmill test) | Within one week before initiating the exercise program
Endurance measure (STEEP treadmill test) | Administered at 6 weeks of the exercise program
Endurance measure (STEEP treadmill test) | Administered at 12 weeks (end of) the exercise program

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Cheifetz O, Dorsay JP, MacDermid JC. Exercise facilitators and barriers following participation in a community-based exercise and education program for cancer survivors. J Exerc Rehabil. 2015 Feb 28;11(1):20-9. doi: 10.12965/jer.150183. eCollection 2015 Feb. PMID 25830140
- [Result] Cheifetz O, Park Dorsay J, Hladysh G, Macdermid J, Serediuk F, Woodhouse LJ. CanWell: meeting the psychosocial and exercise needs of cancer survivors by translating evidence into practice. Psychooncology. 2014 Feb;23(2):204-15. doi: 10.1002/pon.3389. Epub 2013 Sep 6. PMID 24009181